CLINICAL TRIAL: NCT05696821
Title: The POCUS in Practice Study. Implementation of Point-of-care Ultrasonography in General Practice: A Stepped Wedge Cluster Randomized Trial
Brief Title: The POCUS in Practice Study
Acronym: PIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Camilla Aakjær Andersen, Assistant professor, MD, PhD, Aalborg University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Diagnostic
Other Study IDs: ID 242-4
Record Dates: First submitted 2022-09-30; First posted 2023-01-25 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Point-of-care Ultrasound (POCUS)

STUDY DESIGN:
Intervention Model Description: stepped-wedge cluster randomized trial
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the study the intervention cannot be blinded to the participants, but for statistical assessment, data will be blinded as regard to time of collection and location.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Cluster 1 (Other): Participants are randomised into clusters. Each cluster includes 20 participants. All clusters receive the same educational intervention but at different time-points. Each cluster contributes with both exposed and unexposed outcomes and as such acts as its own control.
  Cluster one contributes with 3 months unexposed and 18 months exposed outcomes.
  Interventions: Diagnostic Test: Educational intervention
- Cluster 2 (Other): Participants are randomised into clusters. Each cluster includes 20 participants. All clusters receive the same educational intervention but at different time-points. Each cluster contributes with both exposed and unexposed outcomes and as such acts as its own control.
  Cluster one contributes with 4 months unexposed and 17 months exposed outcomes.
  Interventions: Diagnostic Test: Educational intervention
- Cluster 3 (Other): Participants are randomised into clusters. Each cluster includes 20 participants. All clusters receive the same educational intervention but at different time-points. Each cluster contributes with both exposed and unexposed outcomes and as such acts as its own control.
  Cluster one contributes with 5 months unexposed and 16 months exposed outcomes.
  Interventions: Diagnostic Test: Educational intervention
- Cluster 4 (Other): Participants are randomised into clusters. Each cluster includes 20 participants. All clusters receive the same educational intervention but at different time-points. Each cluster contributes with both exposed and unexposed outcomes and as such acts as its own control.
  Cluster one contributes with 6 months unexposed and 15 months exposed outcomes.
  Interventions: Diagnostic Test: Educational intervention
- Cluster 5 (Other): Participants are randomised into clusters. Each cluster includes 20 participants. All clusters receive the same educational intervention but at different time-points. Each cluster contributes with both exposed and unexposed outcomes and as such acts as its own control.
  Cluster one contributes with 8 months unexposed and 13 months exposed outcomes.
  Interventions: Diagnostic Test: Educational intervention
- Cluster 6 (Other): Participants are randomised into clusters. Each cluster includes 20 participants. All clusters receive the same educational intervention but at different time-points. Each cluster contributes with both exposed and unexposed outcomes and as such acts as its own control.
  Cluster one contributes with 10 months unexposed and 11 months exposed outcomes.
  Interventions: Diagnostic Test: Educational intervention
- Cluster 7 (Other): Participants are randomised into clusters. Each cluster includes 20 participants. All clusters receive the same educational intervention but at different time-points. Each cluster contributes with both exposed and unexposed outcomes and as such acts as its own control.
  Cluster one contributes with 12 months unexposed and 9 months exposed outcomes.
  Interventions: Diagnostic Test: Educational intervention
- Cluster 8 (Other): Participants are randomised into clusters. Each cluster includes 20 participants. All clusters receive the same educational intervention but at different time-points. Each cluster contributes with both exposed and unexposed outcomes and as such acts as its own control.
  Cluster one contributes with 13 months unexposed and 8 months exposed outcomes.
  Interventions: Diagnostic Test: Educational intervention
- Cluster 9 (Other): Participants are randomised into clusters. Each cluster includes 20 participants. All clusters receive the same educational intervention but at different time-points. Each cluster contributes with both exposed and unexposed outcomes and as such acts as its own control.
  Cluster one contributes with 14 months unexposed and 7 months exposed outcomes.
  Interventions: Diagnostic Test: Educational intervention
- Cluster 10 (Other): Participants are randomised into clusters. Each cluster includes 20 participants. All clusters receive the same educational intervention but at different time-points. Each cluster contributes with both exposed and unexposed outcomes and as such acts as its own control.
  Cluster one contributes with 15 months unexposed and 6 months exposed outcomes.
  Interventions: Diagnostic Test: Educational intervention

INTERVENTIONS:
Diagnostic Test: Educational intervention — The educational intervention includes a 3-months training program in the use of point-of-care ultrasound tailored to meet the educational needs of general practitioners. The training programs consists of three teaching seminars over a three month time period, a curriculum of 10 POCUS applications, and an online learning platform providing educational support before, during and after the teaching sessions.

SUMMARY:
In a stepped-wedge cluster randomized trial, the effects of an educational intervention will be determined by estimating the uptake of point-of-care ultrasound by general practitioners (outcome P1), change in referral from primary care to secondary care (outcome P2), change in number of consultations delivered in primary care (outcome S1), GPs job satisfaction, level of stress, and burn-out (outcomes S2-4), as well as the number of point-of-care ultrasound related adverse events (outcome S5), a health economic evaluation (outcome S6) and the patient experience of point-of-care ultrasound (outcome S7).

Two-hundred general practitioners (GPs) will participate in the study. Participants will be randomized to participate in clusters with a training facility close to their clinic. All participants will be offered the educational intervention. Ten clusters will receive the intervention at different timepoints.

DETAILED DESCRIPTION:
In a stepped-wedge cluster randomized trial the effects of an educational intervention, where general practitioners (GPs) are trainined in the use of point-of-care ultrasound (POCUS) in office-based general practice, will be dertermined.

The intervention is in line with international recommendations for ultrasound education and consists of three teaching seminars over a three month time period, a curriculum of 10 POCUS applications, and an online learning platform providing educational support before, during and after the teaching sessions.

The online platform includes instruction videos demonstrating the performance of POCUS, assignments to support the development of skills, self-tests to focus attention of learning outcomes and specific actioncards for each of the 10 POCUS applications framing the examinations in the clinical context. In addition, the online platform gives participants access to webinars and communication with other participants and teachers, who will act as mentors during the learning process.

Two-hundred GPs will participate in the study. Participants will be randomized to participate in clusters. Ten clusters will receive the educational intervention at different timepoints. Each cluster will consists of a group of 20 GPs from the same geographical area (the five Danish regions).Hence, the study will include two clusters from each of the five Danish regions, who will receive the educational intervention at a location in the specific region ( Copenhagen, Lyngby, Roskilde, Næstved, Odense, Vejle, Aarhus, Herning, Sæby and Aalborg) at different timepoints.

Participants Recruitment All GPs working in Danish general practice will be invited to participate in the study by an e-mail circulated by the Organisation of General Practitioners in Denmark (Praktiserende Lægers Organisation - PLO) to all PLO members. The e-mail will contain a link to a questionnaire in which the GPs will be asked to specify their name, practice, location of practice (region in Denmark), distance to nearest ultrasound scanning service, whether or not they are already using POCUS, whether or not they will have access to an ultrasound device during the educational intervention, and whether or not they are willing to share data. There will be a deadline for responding to the invitation.

Eligibility criteria for participation Following the deadline for signing up to participate in the study, the GPs reply to the questionnaires will be screened according to the inclusion and exclusion criteria to make a list of eligible participants fulfilling all inclusion and none of the exclusion criteria.

Selection of participants The selection of participants follows the below prioritizing.

1. The list of eligible participants will be sorted based on geography (based on regions) and according to the GPs distance to the nearest ultrasound scanning service. In each region, the 40 GPs with the longest distance to an ultrasound scanning service, will be offered to participate in the study.
2. In case a GP, offered to participate in the study, does not wish to participate, the offer will be given to the next on the list.
3. In case there are less than 40 participants in a region, eligible GPs from the neighbouring region with the longest distance to an ultrasound scanning service, will be allocated to the region with less than 40 participants.
4. POCUS-users account for approximately 12% of all PLO members (unpublished data). Therefore, only approximately 12% (five GPs per region) of eligible participants can be POCUS-users. If the prioritized list includes more than five POCUS-users, the first five POCUS-users on the list will be considered and the remaining POCUS-users will be excluded giving way for non-users further down the list to be considered.

Hence, the final list of eligible GPs, who will be offered participation in the studies, will include 200 GPs, with a maximum of 25 POCUS-users, working in the general practice clinics with the longest distance to ultrasound scanning services.

In case all non-users on the prioritized list have been offered to participate in the study, and some does not wish to participate, the remaining openings will be offered to eligible POCUS users - giving way for more than 25 POCUS-users to be included in the study.

Allocation When the GPs sign up to participate in the study, they will be able to see the participation dates at each training facility (Copenhagen, Lyngby, Roskilde, Næstved, Odense, Vejle, Aarhus, Herning, Sæby and Aalborg). Each region offers two sets of dates. The GPs will know the two sets of dates in their region, but not which one their will be allocated to (this will be determined on behalf of randomization).

Once 200 GP have been allocated to the five training facilities used in the SW-CRT, the 40 participants allocated to each region will be randomized to participate in one of the two clusters (group of GPs receiving the intervention at a given location and time period).

Randomisation Randomisation will be performed on two levels - cluster order and individual participation at a specific time.

Order of clusters First, the overall order of all clusters will be randomized. I.e. the order of the clusters defined by each location are decided based on simple randomization -drawing an anonymous paper slip at random order with one of the following texts: Copenhagen, Lyngby, Roskilde, Næstved, Odense, Vejle, Aarhus, Herning, Sæby and Aalborg. From this an order for the delivery of courses is established. This randomisation and the fixed timeline for the delivery of these courses will be done on June 17th 2022 in order to plan and prepare the delivery of the intervention.

Participants' time of intervention The randomisation of participants at a given location to receive the intervention at one of two time points of will take place after the deadline for signing up for the course prior to the start of the data collection. The randomisations will be done by a research assistant not involved in assessment or delivery of the intervention. The randomization process will be video documented.

Following this randomization process, the GPs will be offered participation in the SW-CRT by e-mail including a link for the PLO-e course allocated to the specific cluster.

Outcomes and data

Registry data:

Following the use of POCUS in the general practice consultations the GPs will follow normal procedures for registration of activities in general practice using remuneration codes, fee-specific codes for using POCUS, and referrals in the medical record system. Prior to this study 11 fee-specific codes for 11 different POCUS examinations will be installed in the medical record system. The Primary Sector Data Provider Platform (PLSP) will develop an algorithm that allows for the following data extraction on each participating GP in a given time frame: (1) number of POCUS examinations performed, (2) number of referrals, and (3) number of consultations (outcomes P1, P2, S1 and S5). PLSP will deliver monthly aggregated data for each participating GP.

General practitioner data:

For the GP questionnaire (outcomes S2-S4), validated scales will be used to determine GPs' perceived stress (Cohen's 10-item Perceived Stress Scale), GPs' job satisfaction (Warr-Cook-Wall Job satisfaction Scale) and GPs burnout symptoms (Maslach Burnout inventory). Prior to the study, these questionnaires were tested for face validity in four focus groups with 18 POCUS using GPs (unpublished materiel). The Cohen's 10-item Perceived Stress Scale includes ten items about the frequency of stress-related feelings and thoughts. Each item is rated from 0 (never) to 4 (very often). Previous research has reported a sum score of ≥ 18 to be a high level of stress . The Warr-Cook-Wall Job satisfaction Scale includes 9 sub-items measuring facets of job satisfaction and one overall item rated on a scale from 1 (extreme dissatisfaction) to 7 (extreme satisfaction). In previous research25 a cut-off on the overall item of ≤ 3 has been used to identify low job satisfaction. The Maslach Burnout inventory consists of 22 items exploring the following three burnout dimensions: (1) emotional exhaustion (9 items) characterised by depletion of emotional resources, (2) depersonalisation (5 items) characterised by emotional detachment from people related to work including patients and (3) personal accomplishment (8 items) including perceived value of work and self-efficacy. All dimensions are rated on a scale from 0 (never) to 6 (every day). A sum score is calculated for each dimension. For each scale, a mean sum score with SD and a median sum score with IQR will be calculated.

For the tertiary outcomes T1-T3, items previously developed and validated in Danish general practice will be used measuring aspects of GP's job contentment (T1), GPs' experience of POCUS use in general practice (T2) and finally, the GPs will be asked to declare on a 5-point-likerts scale if they agree or disagree that POCUS use had influenced their sense of perceived stress, job satisfaction or burnout symptoms (T3).

Patient data: (outcome S6) A patient questionnaire will be delivered to all patients (≥ 18 years old) examined with POCUS, who will be able to provide an informed consent, in month 5-6 after the educational intervention. Patients will fill out the questionnaires themselves using their own mobile devices. The questionnaire will be accessed using GP specific QR-codes (or alternatively a paper questionnaire). Items previously developed and validated will be used (see the attached study protocol).

Possible adverse events: (outcome S7) For the registration of possible adverse events, a questionnaire will be used giving the GPs the possibility to explain in free text using their own words to explain (1) what was scanned, (2) circumstances surrounding the scan, (3) what happened, and (4) reflections after the scan. This reporting of cases will be anonymous. Data will be collected from the educational intervention to the end of the study. The aggregated total number of monthly registrations for each participating GP will be reported.

Evaluation of the patient pathway and quality of selected POCUS examinations: (outcome S8) After the study, participating GPs will be instructed to make an evaluation of the patient pathway following selected POCUS examinations. A separate protocol will be developed for this part.

Background characteristics of participating GPs At baseline the following participant characteristics will be collected in a baseline questionnaire: Age (years), gender (M, F, other), seniority (year of graduation from medical school), experience (years working as a GP), previous use of ultrasound (number of years with regular use), previous ultrasound training (yes,no), scanner type (low range, mid range, high end), practice owner (yes, no), type of practice (collaboration, partnership, solo), location of practice (urban, rural, mixed), distance to the nearest imaging facility, number of patients assigned to the practice, and number of GPs working in the practice. In addition, the GP's participation in educational activities during the educational intervention will be registrered.

Characteristics of scanned patients From PLSP, aggregated data (age, gender) on patients will be received. Patients, who have had a POCUS fee-specific code registered in their medical record during the study.

The data management will follow the rules of the General Data Protection Regulaton (GDPR) and the Danish Data Protection Agency (registration number 2022-068-03601). All study data will be stored on a secure server at Aalborg University.

Sample size This is a pragmatic trial where size of the sample is given by the collectice agreement between PLO and the Danish Regions. Post-hoc power calculations to support the reliability of analytic findings are planned.

Statistical methods All statistical analyses will be performed using STATA version 17 (StataCorp, Texas, USA).

The principles of Intention-to-treat is followed in the analysis. If a GP e.g. misses one teaching seminar, the GP is still considered has having completed the educational intervention. Data will be analyzed according to a pre-established Statistical Analysis Plan (SAP) in consultation with a statistician. For the primary outcomes (continuous data), linear regression models adjusting for the fixed effect of time and the random effects of clusters are planned.

Due to the nature of the study the intervention cannot be blinded to the participants, but for statistical assessment, data will be blinded as regard to time of collection and location.

Ethics and conflicts of interests The study will be performed in accordance with the Declaration of Helsinki. The project was notified to the regional ethical committee (The North Denmark Region Committee on Health Research Ethics, registration number 96036), who responded that do ethical approval was necessary. The trial may be discontinued for a patient, a GP, a general practice clinic, and a cluster in case of withdrawal of an informed consent.

External sponsors have no part in the study design, data analyses or writing of the manuscript. The authors declare no conflict of interest.

ELIGIBILITY:
Inclusion criteria:

1. GPs who are postgraduate medical doctor with a specialization in general practice
2. GPs who work in office-based Danish general practice
3. GPs who have access to an ultrasound device in the practice during the study period

Exclusion criteria:

1. GPs not willing to participate in the data collection or share data for this study
2. No signed informed consent to participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
The uptake of the intervention in primary care | months 3- 21
  The effect on the uptake of POCUS following an educational intervention for general practice clinics will be determined by comparing the number of registered reimbursement codes before the intervention to the number of reimbursement codes registered after the intervention.
Change in number of referrals for secondary care | months 1- 21
  The effects of an educational intervention for general practice clinics on the number of referrals send to secondary care specialists, will be determined by comparing the number of registered referrels (number of referrals to hospital or specialist clinics/number of consultations) before the intervention to the number of registered referrals after the intervention.

SECONDARY OUTCOMES:
Change in number of consultations in primary care | months 1- 21
  The effects of an educational intervention for general practice clinics on the number of consultations in general practice, will be determined by comparing the number of registred consultations (e-mail, telephone, video, GP office, visits) before the intervention to the number of registered consultations after the intervention.
Change in GPs' perceived stress | Estimated in each cluster 1 months before the intervention and six months after the intervention
  The effects of an educational intervention on GPs' perceived stress, will be measured by comparing Cohen's 10-item Perceived Stress Scale before and after the educational intervention.
Change in GPs' job satisfaction | Estimated in each cluster 1 months before the intervention and six months after the intervention
  The effects of an educational intervention on GPs' job satisfaction, will be measured by comparing Warr-Cook-Wall Job satisfaction Scale before and after the educational intervention.
Change in GPs' burnout symptoms | Estimated in each cluster 1 months before the intervention and six months after the intervention
  The effects of an educational intervention on GPs' burnout symptoms, will be measured by comparing Maslach Burnout inventory before and after the educational intervention.
Change in healthcare costs | months 1-21
  The effects of an educational intervention on healthcare costs, will be measured by comparing costs before and after the educational intervention.
Patient experience | In each cluster months 5-6 after the intervention
  The patient experience following the educational intervention, will be determined using patient questionnaires following the intervention
Possible adverse events | months 1-21
  The number of self-reported POCUS-related possible adverse events following the educational intervention, will be determined using questionnaires for the participating GPs.

OTHER OUTCOMES:
Change in GPs' job contentment | Estimated in each cluster 1 months before the intervention and six months after the intervention
  GPs' experiences of job contentment will be measured using specific items in a questionnaire before and after the intervention
GPs' experience of POCUS use | Estimated in each cluster six months after the intervention
  GPs' experience of POCUS use in their practice, will be measured using specific items in a questionnaire after the intervention
GPs' experiences of POCUS' influence | Estimated in each cluster six months after the intervention
  GPs' experiences of POCUS' influence on perceived stress, job satisfaction and burnout symptoms will be measured using specific items in a questionnaire after the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Center for General Practice at Aalborg University, Aalborg, Denmark

DOCUMENTS (2):
  • Study Protocol (2022-12-27): https://cdn.clinicaltrials.gov/large-docs/21/NCT05696821/Prot_001.pdf
  • Statistical Analysis Plan (2024-12-19): https://cdn.clinicaltrials.gov/large-docs/21/NCT05696821/SAP_002.pdf